CLINICAL TRIAL: NCT01656694
Title: Two and Five-Year Survivorship of Unicompartmental Knee Arthroplasty Using DePuy Sigma HP Replacement
Brief Title: A Single-Center, Epidemiological Study of the Survivorship of the DePuy Sigma HP Unicompartmental Knee Prosthesis
Status: Completed | Type: Observational
Sponsor: Mississippi Sports Medicine and Orthopaedic Center (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Other Study IDs: 11018
Record Dates: First submitted 2012-08-01; First posted 2012-08-03 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Osteoarthritis; Unicompartmental Knee Arthroscopy
Keywords: Osteoarthritis; Knee; Replacement; Unicompartmental; DePuy; Sigma HP
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: DePuy Sigma HP Partial Knee

SUMMARY:
This study will be conducted to assess the survivorship of a particular prosthesis used in unicompartmental knee arthroplasties. Patients undergoing this procedure have been diagnosed with isolated medial or lateral compartmental arthritis and have failed conservative treatment. The patients received a unicompartmental knee replacement using the Sigma® HP Partial Knee System.

DETAILED DESCRIPTION:
This study is an epidemiological Level IV-Case Series clinical study that will study the survivorship of the Sigma® HP Partial Knee System in a consecutive series of patients. All patients who received the Sigma® HP Partial Knee System between August 21, 2008 and October 31, 2009 will be available to include in the study. Data will be collected preoperatively, intra-operatively, and post-operatively at intervals of 6 weeks, 6 months, 1 year, 2 years, and 5 years. Data will be analyzed for survivorship status at the 2- and 5-year follow-up visits. Other data, including functional outcomes, radiographic outcomes, and wear will be analyzed at the 5-year follow-up visit. Subjects will participate in the study for five years after their surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient over the age of 18
* Diagnosis of isolated medial or lateral compartmental osteoarthritis of the knee joint
* Must have failed conservative treatment and received a unicompartmental knee arthroplasty between August 21, 2008 and October 31, 2009.
* Must have received the Sigma® HP Partial Knee System.
* Must have received the surgery from Dr. Almand, Dr. Johnson, or Dr. Pickering at Mississippi Sports Medicine and Orthopaedic Center.
* Must be willing to provide written consent to participate in the study.
* Subjects who do not have the legal capacity to consent may be enrolled in the study by a Legally Authorized Representative (LAR). The LAR must provide verification that they have the legal authority to represent the subject.

Exclusion Criteria:

* Did not receive a unicompartmental knee arthroplasty between August 21, 2008 and October 31, 2009.
* Did not receive a unicompartmental knee arthroplasty using the Sigma® HP Partial Knee.
* Did not receive their unicompartmental knee replacement from Dr. Almand, Dr. Johnson, or Dr. Pickering at Mississippi Sports Medicine and Orthopaedic Center.
* Subjects lost to follow-up for any reason including, but not limited to: refusal to consent, death, or geographic isolation will also be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Since the first Sigma® HP Partial Knee System was introduced at MSMOC, over 1,000 have been implanted in patients by the investigators of this study. The population used for this study was the first patients of our clinic to receive this particular prosthesis. The first replacement was implanted on August 21, 2008. By October 31, 2009, 300 patients had received the Sigma® HP replacement. These 300 patients will be the subject population whose data will be analyzed for the study upon their consent.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2012-08; Primary Completion 2015-12-31 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Five-Year Survivorship | Five Years Post-Op
  The primary endpoint of the study is to determine the five-year survivorship of the Sigma® HP Partial Knee System with failure defined as revision for any reason.

SECONDARY OUTCOMES:
Five-Year Survivorship Alternately Defining Failure and Two-Year Survivorship | Two Years and Five Years Post-Op
  One secondary endpoint of the study is to determine the five-year survivorship of the prosthesis with alternately defining failure as: failure of implant, failure secondary to infection, failure secondary to progression of arthritis, failure secondary to periprosthetic fracture.
  We also want to determine the two-year survivorship with failure defined as revision for any reason.
Functional Outcomes | Five Years Post-Op
  Another secondary endpoint of the study is to analyze the functional outcomes for five-year data based on the Knee Society score and the KOOS (Knee Injury and Osteoarthritis Outcome Score) score, reported as changes from the pre-operative score. By using both rating systems, an appropriate evaluation of the functional outcome of the surgery should be obtained.
Radiographic Outcomes | Pre-Operatively, Two and Five-Year Post-Op
  Another secondary endpoint of the study is to determine the radiographic outcomes based upon the radiographic assessment using the Knee Society scoring system, reported as changes from the pre-operative assessment. Additionally, we want to radiographically assess lucencies at the bone cement and implant cement interface to measure wear and loosening of the prosthesis.
Adverse Advents | Post-Operatively
  We also want to examine the type and frequency of adverse events as a secondary endpoint of the study. Safety will be evaluated with summary of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff D Almand, MD, Principal Investigator — Mississippi Sports Medicine and Orthopaedic Center
Locations (1):
- Mississippi Sports Medicine and Orthopaedic Center, Jackson, Mississippi, United States